CLINICAL TRIAL: NCT02760979
Title: The Efficacy of Denosumab in Decreasing Periprosthetic Bone Loss in Patients With Total Knee Arthroplasty: A Randomised, Double Blind, Placebo Controlled Clinical Trial
Brief Title: The Efficacy of Denosumab in Decreasing Periprosthetic Bone Loss in Patients With Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IIBSP-DEN-2012-24; 2012-001285-15 (EudraCT Number)
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Bone Resorption
Keywords: knee arthroplasty
MeSH Terms: conditions — Bone Resorption | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denosumab (Active Comparator): Patients treated with Denosumab
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): Patients treated with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denosumab — Denosumab treatment one year after surgery
  Other Names: Prolia
  Arms: Denosumab
Drug: Placebo — Serum one year after surgery
  Other Names: Serum
  Arms: Placebo

SUMMARY:
This study evaluates the effect of Denosumab in decreasing the periprosthetic bone resorption after Total Knee Arthroplasty compared to placebo in 60 patients (30 placebo and 30 Denosumab) within a year after surgery.

DETAILED DESCRIPTION:
Periprosthetic bone resorption after Total Knee Arthroplasty occurs as a consequence of prosthetic implant on the bone. Some of this patients (up to 13%) develop an aseptic failure of the prosthesis needing revision surgery.

2 groups of patients are treated with Placebo and Denosumab in a double blind prospective trial. Densitometry, Knee society score (KSS), Western Ontario McMaster University Osteoarthritis Index (WOMAC) and the Medical Outcomes Study Short Form 36 (SF-36) were done in both groups at 0,3,6 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Knee Osteoarthritis treated with Total Knee Arthroplasty

Exclusion Criteria:

* Patients allergies to Denosumab
* Patients with previous Osteoporosis treatment
* Patients with renal failure
* Patients with previous Bisphosphonate treatment for more than 5 years

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Bone Mass index | Change in densitometry before surgery (0) and at three (3) months after surgery
  Bone Mass index in gr/cm3
Change in Bone Mass index | Change in densitometry before surgery (0) and at six (6) months after surgery
  Bone Mass index in gr/cm3
Change in Bone Mass index | Change in densitometry before surgery (0) and at twelve (12) months after surgery
  Bone Mass index in gr/cm3

SECONDARY OUTCOMES:
Quality of Life (WOMAC) | WOMAC test before (0) and at three (3), six (6) and twelve (12) months after surgery
Quality of life (SF-36) | SF-36 test before (0) and at three (3), six (6) and twelve (12) months after surgery
Kidney function | Before surgery and at three, six and twelve months after surgery
  Creatinine clearance
Liver function | Before surgery and at three, six and twelve months after surgery
  ALT, AST
Bone turnover markers | At three, six and twelve months after surgery
  Beta cross lap and Procollagen type 1 n-terminal propeptide (P1NP)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos Gonzalez, Principal Investigator — Orthopaedic Department-Hospital de la Santa Creu i Sant Pau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishii Y, Yagisawa K, Ikezawa Y. Changes in bone mineral density of the proximal femur after total knee arthroplasty. J Arthroplasty. 2000 Jun;15(4):519-22. doi: 10.1054/arth.2000.4639. PMID 10884214
- [Background] Sugita T, Umehara J, Sato K, Inoue H. Influence of tibial bone quality on loosening of the tibial component in total knee arthroplasty for rheumatoid arthritis: long-term results. Orthopedics. 1999 Feb;22(2):213-5. doi: 10.3928/0147-7447-19990201-10. PMID 10037335
- [Background] Wang CJ, Wang JW, Weng LH, Hsu CC, Huang CC, Chen HS. The effect of alendronate on bone mineral density in the distal part of the femur and proximal part of the tibia after total knee arthroplasty. J Bone Joint Surg Am. 2003 Nov;85(11):2121-6. doi: 10.2106/00004623-200311000-00009. PMID 14630840